CLINICAL TRIAL: NCT02953366
Title: Phase III, National, Multicenter, Randomized, Single-blind, Non-inferiority to Compare the Efficacy of Mometasone Nasal Gel Compared to Mometasone Nasal Spray in the Treatment of Persistent or Intermittent Allergic Rhinitis in Childrens
Brief Title: Efficacy and Safety of the Mometasone Nasal Gel in the Treatment of Persistent Allergic Rhinitis
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: EMS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EMS1215
Record Dates: First submitted 2016-11-01; First posted 2016-11-02 (Estimated); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic | interventions — Mometasone Furoate

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EMS Mometasone gel (Experimental): The patient should administer 1 spray in each nostril once daily.
  Interventions: Drug: EMS Mometasone gel
- Mometasone spray nasal (Active Comparator): The patient should administer 1 spray in each nostril once daily.
  Interventions: Drug: Mometasone spray nasal

INTERVENTIONS:
Drug: EMS Mometasone gel — The patient should administer 1 spray in each nostril once daily.
  Arms: EMS Mometasone gel
Drug: Mometasone spray nasal — The patient should administer 1 spray in each nostril once daily.
  Other Names: Nasonex
  Arms: Mometasone spray nasal

SUMMARY:
The purpose of this study is to evaluate the non-inferiority of the clinical efficacy of the mometasone nasal gel in the treatment of allergic rhinitis.

ELIGIBILITY:
Inclusion Criteria:

* Signed Consent of the patient;
* Clinical diagnosis of moderate - severe persistent allergic rhinitis according to ARIA classification(Allergic Rhinitis and Its Impact on Asthma);

Exclusion Criteria:

* Patients with any clinically significant disease that in the investigator is opinion can´t participate in the study;
* Patients with any laboratory finding or image finding that in the investigator is opinion can´t participate in the clinical trial;
* Patients with history of hypersensitivity to any of the formula compounds;
* Participation in clinical trial in the year prior to this study;
* Pregnancy or risk of pregnancy and lactating patients;
* Patients who were in use of drugs that can interfere with evaluation;
* Decongestants dependent patients or patients receiving allergen specific immunotherapy;
* Patients on treatment with monoamine oxidase inhibitors (MAOIs).

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2019-05 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Efficacy of allergic rhinitis treatment based proportion of participants who show at least moderate relief. | 28 days

SECONDARY OUTCOMES:
Safety will be evaluated by the adverse events occurrences | 28 days